CLINICAL TRIAL: NCT02862002
Title: Measuring the Effects of Therapeutic Education Program "Caratif" Patient Under Strong Opioids Versus Standard Taking Charge of Patient Pain Receiving Opioid Therapy in Medical Oncology.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: RC12_3975 - 2756
Record Dates: First submitted 2016-08-05; First posted 2016-08-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Pain Management
Keywords: opioid therapy; medical oncology.
MeSH Terms: conditions — Agnosia | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapeutic Patient Education (E.T.P)of type "caratif (Experimental): Patients in arm E.T.P benefit of the nursing consultation E.T.P,
  Interventions: Other: therapeutic education of type "caratif; Other: Standard care
- standard care (Active Comparator): patients receiving standard care of cancer pain.
  Interventions: Other: therapeutic education of type "caratif; Other: Standard care

INTERVENTIONS:
Other: therapeutic education of type "caratif — study the effects of a therapeutic education program type "caratif", based on a communication pedagogy, with the patient receiving opioid therapy in medical oncology
Other: Standard care — patients receiving standard care of cancer pain.

SUMMARY:
A first empirical evidence on the difficulties of observance of morphine in cancer patients invited a multidisciplinary team to initiate an innovative quality approach. It shows the lack of transcript of a comprehensive care causing a problem for monitoring actions undertaken for the relief of pain. In addition, two exploratory studies targeting the expectations and needs of the Patient Therapeutic Education (E.T.P) receiving strong opioids.

The E.T.P, public health priority, provides a framework for action and improving care. In oncology, the involvement of the patient in pain relief and management of opioids represents an axis of intervention more appropriate. Yet, it is not found in literature. In our department, we conduct an experimental therapeutic education program type "caratif" and a nurse consultation FTE receiving opioids on the model of nursing "care" of J. Watson (humanist emphasis promoting interpersonal teaching-learning mobilizing the patient experience). The ETP folder and its tools have been continuously validated with patients. The heart of the educational process is in the patient's complex path neat oncology and relies on interaction and creativity between patient and caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Cancer patients receiving opioids
* Suffering from pain caused by their disease or treatment with chemotherapy and / or radiotherapy and / or surgery
* Supported within the oncology or palliative care
* Receiving at least 3 courses of chemotherapy
* Having read, understood and signed the informed consent
* Subject beneficiary of a social security scheme or an equivalent -

Exclusion Criteria:

* adults subject to a legal protection measure or unable to consent
* Non-beneficiaries of a social security scheme,
* persons deprived of liberty by a judicial or administrative decision,
* patients with neurological or psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Pain assessment | 21 days
  Using a digital scale

SECONDARY OUTCOMES:
Treatment adherence morphine | 21 days
  Digital Scale / self-administered questionnaire of adherence of Girerd et al [78]
Strategies Adjustment disease | 21 days
  Scale MAC (Mental Adjustment to Cancer Scale) French Version: Cayrou et al, 2001 [82]
Anxiety | 21 days
  Scale HADS (Hospital anxiety and depression seale, French version: Sigmund and Snaith) [83]
Depression | 21 days
  Scale HADS (Hospital anxiety and depression seale, French version: Sigmund and Snaith) [83]

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille Hôpital de la Timone, Marseille, France